CLINICAL TRIAL: NCT02070276
Title: Can Non Invasive Methods for Fluid Responsive Assessment Optimize Preventive Volemic Repletion in Order to Prevent Significant Hypotension After Spinal Anesthesia? A Randomized Trial
Brief Title: Predict Fluid Responsiveness in Spinal Anesthesia
Acronym: CERU-1401
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Principal Investigator, Samuele Ceruti, Capoclinica Medicina Intensiva, Ente Ospedaliero Cantonale, Bellinzona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CERU-1401; ProCRHYSA trial (Other Grant/Funding Number: ABREOC)
Record Dates: First submitted 2014-02-18; First posted 2014-02-25 (Estimated); Results first posted 2019-12-19 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Hypotension and Shock; Excessive Amount of Blood / Fluid Infusion
Keywords: Fluid therapy; Hypotension; Inferior vein cava; Spinal anesthesia; Ultrasonography
MeSH Terms: conditions — Hypotension; Shock

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Clinical Practice (No Intervention): This arm is considered the current clinical standard for spinal anesthesia; its used as a control sample and statistical reference. During the induction phase the patient is fitted with a non-invasive blood pressure monitoring, three-lead ECG, pulse oximetry and peripheral intravenous device. The pressure control is set as the standard every 5 minutes until the procedure under spinal anesthesia, the cuff pressure is placed on the arm that is going to be on top during spinal anesthesia.
  Data is recorded and vital signs of the patient and is put an infusion of crystalloid (0.9% NaCl or Ringer's acetate) with administration of 500 ml during the entire procedure until the beginning of the operation.
- Trans-thoracic echocardiography (Experimental): In addition to the current clinical standard (arm A of the study) a trans-thoracic echocardiography is performed with the aim of assessing patient's volume status, identifying if he is responsive to fluid and could benefit from their administration. The echocardiography is performed with the subcostal projection to assess the size of the abdominal inferior vena cava and its collapsing during breathing.
  According to different pre-established parameters, the patient is defined as unresponsive to fluids or responsive. If it's not responsive, he proceed to spinal anesthesia. Otherwise investigators proceed to the administration of crystalloid (NaCl 0.9% or Hartmann's solution second clinical evaluation) and at the end he's rerun an echocardiographic assessment.
  Interventions: Procedure: Trans-thoracic echocardiography
- Passive Leg Raising Test (Experimental): In addition to the arm A of the study, is performed a measurement of end-tidal CO2 (EtCO2) by trans-nasal canula with a patient positioned in semi-recumbent position. After, investigators run the Passive Leg Raising Test (PLRT): the position of the bed is changed in such manner to bring the trunk from 45° to 0° and accordingly the legs from 0° to 45°. Measurements are performed before and during the maneuver : an etCO2 increasing more than 12% from baseline was interpreted as fluid-responsive.
  If the patient is not responsive to fluids, the patient is moving to the spinal anesthesia. If the patient is responsive investigators proceed to bolus administration, the patient returns to the initial PLRT position and is run again the PLRT until the patient is no longer responsive to fluids.
  Interventions: Procedure: Passive Leg Raising Test

INTERVENTIONS:
Procedure: Trans-thoracic echocardiography — Subcostal evaluation of inferior vena cava dimensions and colorability with cyclic spontaneous breathing in order to determine if the patients will be fluid responsive or not.
  Arms: Trans-thoracic echocardiography
Procedure: Passive Leg Raising Test — Application of this test in a standard manner in order to determine if our spontaneous breathing patients are fluid responsive before spinal anesthesia.
  Arms: Passive Leg Raising Test

SUMMARY:
Spinal anesthesia is still the regional anesthesia technique most widely employed in everyday clinical practice.

The most feared and common of its well known side effects consist in an abrupt reduction of systemic vascular resistances, with consequence risk of systemic hypotension. To prevent this potentially severe complication, an adequate correction of patients' volume status through a preventive administration of fluids is widely used.

However this volume repletion is commonly accomplished on an empirical basis, without having a real insight of patient hemodynamic status, carrying the risk of possible volume overload.

Aim of the study is to test the clinical impact of two simple, non-invasive methods to guide volemic repletion before spinal anesthesia on the reduction of significant hypotension rate, compared to empirical fluid administration.

DETAILED DESCRIPTION:
The resulting high density of the anesthetic block and the reproducibility of the technique have made of spinal anesthesia the most widely diffused regional anesthesia technique. Nevertheless the procedure still remains the regional anesthesia technique burdened by the potentially most severe side effects, the most frequent of which being systemic arterial hypotension.

Subarachnoidal administration of local anesthetics in fact is associated not only with both a motor and sensory block, but also with a blockade of the autonomic nervous system, which controls peripheral vascular tone. Sympathetic block leads to a sudden decrease in peripheral resistance, with consequent significant increase in vascular bed and relative hypovolemia.

Transient hypotensive episodes can be generally well tolerated by healthy patients, however they may lead to major complications in patients with increased cardiovascular risk. In the common clinical practice, it is usual to administer fluids empirically. An empirical preventive fluid repletion however can represent per se a risk in patients with impaired cardiac and renal functions, since a volume overload of heart chambers with reduced compliance can cause pulmonary edema or congestive heart failure.

Since about ten years both non-invasive and invasive techniques have been developed, with the specific purpose of optimizing fluid status on a rational basis. This methods are based on the correlation between the levels of mean arterial pressure (MAP), systemic vascular resistance (SVR) and cardiac output (CO), according to the equation: MAP = CO * SVR. The latter explains why, in case of vasodilation, unless CO is increased, a lowering of SVR will inevitably translate into a decrease of MAP.

Determinants of blood pressure are:

1. volemic status;
2. vascular resistance (determined by the control of the sympathetic system);
3. cardiac output.

In case of spinal anesthesia the reduction in SVR determines relative hypovolemia (due to an increase in total vascular bed). For this reason after spinal anesthesia appears fundamental an optimization of patients' volemic status through administration of fluids (eventually associated with the administration of amines, in order to contrast massive vasodilation).

The use of methods to assess fluid responsiveness has been extensively studied in critical patients populations. However these techniques have not been studied yet in non critical patients. Spinal anesthesia is a model of pharmacological vasodilation which often generates significant hypotension, for which nowadays an evidence-based rational treatment based on a guided volemic repletion is still lacking.

WORKING HYPOTHESIS:

The use of non-invasive methods that have proven to be accurate for the identification of patient fluid-responsiveness is currently not validated in patients undergoing spinal anesthesia.

Ultrasound of inferior vena cava by is an effective method to determine the responsiveness to fluids in a patient on mechanical ventilation, however it has been proven to be inaccurate in spontaneous ventilating patients in critically ill patients, few data being available in non critical patients. The study of the inferior vena cava is based on the size of the inferior vena cava in its intra-abdominal portion (approximately 2 cm from emergency right atrium) and the pattern of its diameter changes with breathing. This measurement is obtained with M-mode ultrasound through subcostal view..

Passive leg raising test (PLRT) has been proven to be a highly accurate method in predicting fluid responsiveness in spontaneously breathing patients, in a population of critically ill patients. The method is based on the following assumption: active legs elevation, in addition to its effect of venous pool shifting from the lower limbs to the thorax, exerts a contemporary effect of stimulation on the peri-arterial sympathetic system at iliac-femoral level, this causing an orthosympathetic reflex which can increase cardiac output, possibly masking hypovolemia. Passive lower limbs raising instead has the advantage of mobilizing lower limbs venous blood (estimated 300-500 ml), without activating the orthosympathetic reflex. This allows for a quantification of the clinical response to a bolus of fluids, in terms of decrease of blood pressure variations following leg raising.

The hypothesis that investigators want to test is that the use of inferior vena cava ultrasound before spinal anesthesia, compared to the standard method (empirical fluid administration) and a non-invasive method (PLRT) can reduce the impact of systemic hypotension through an adequate titrated volemic repletion, avoiding both hypotension and fluid overload. The final purpose is to ensure spinal anesthesia in the safest possible way.

OBJECTIVES OF THE STUDY:

Aim of the study is to determine whether vena cava ultrasound, a bedside, unexpensive, non invasive methods, which have been tested as predictors of fluid responsiveness in critical patients, is effective in guiding titrated fluid repletion in a non critical population, in order both to decrease post procedural significant hypotension rate and unnecessary fluid overload in patients undergoing spinal anesthesia for elective surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* all adult non critical patients requiring elective spinal anesthesia
* both sex
* patients with American Society of Anesthesiology class level I, II and III according to international standards
* spontaneously breathing patients

Exclusion Criteria:

* patients already equipped or requiring invasive blood pressure monitoring (arterial catheter, pulmonary catheter, thermodilution catheter)
* patients with pre-procedural hypotension, defined as a response in two consecutive measurements of systolic arterial pressure (SAP) less than 80 mmHg or mean arterial pressure (MAP) less of 60 mmHg.
* patients unable to give informed consent to communication difficulties to language barriers or processes congenital/acquired determinants of mental retard, or any reduction in their ability to understand or want to be able to give their informed consent to the study
* patients where it is not then possible to perform spinal anesthesia for the patient's refusal to technical difficulties in sampling, clinical pathological conditions for determining a high risk of peri- procedural complications.
* patients with International Normalized Ratio > 1.5 and/or activated partial thromboplastin time in therapeutic range (defined as a value more than 1.5-2 times the normal values of the patient), anti-Xa activity in the therapeutic range .
* patients with severe thrombocytopenia (<50 G/l)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2014-05; Primary Completion 2019-02 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuele Ceruti, MD, Principal Investigator — Ente Ospedaliero Cantonale - Ospedale Regionale di Bellinzona; Andrea Saporito, MD, Study Chair — Ente Ospedaliero Cantonale - Ospedale Regionale di Bellinzona
Locations (1):
- Ospedale Regionale di Bellinzona e Valli (ORBV) - Sede Bellinzona, Bellinzona, Switzerland

REFERENCES:
- [Background] Kim HJ, Kim JS. A cardiovascular collapse following vigorous cough during spinal anesthesia. Korean J Anesthesiol. 2013 Dec;65(6 Suppl):S49-50. doi: 10.4097/kjae.2013.65.6S.S49. No abstract available. PMID 24478870
- [Background] Nogueira CS, Lima LC, Paris VC, Neiva PM, Otani ET, Couceiro Rde O, Burim F, Ferreira JA Jr, Cadecaro P. A comparative study between bupivacaine (S75-R25) and ropivacaine in spinal anesthesia for labor analgesia. Rev Bras Anestesiol. 2010 Sep-Oct;60(5):484-94. doi: 10.1016/S0034-7094(10)70060-X. English, Portuguese. PMID 20863929
- [Background] Xu S, Wu H, Zhao Q, Shen X, Guo X, Wang F. The median effective volume of crystalloid in preventing hypotension in patients undergoing cesarean delivery with spinal anesthesia. Rev Bras Anestesiol. 2012 May-Jun;62(3):312-24. doi: 10.1016/S0034-7094(12)70132-0. PMID 22656677
- [Background] Kaimar P, Sanji N, Upadya M, Mohammed KR. A comparison of hypotension and bradycardia following spinal anesthesia in patients on calcium channel blockers and beta-blockers. Indian J Pharmacol. 2012 Mar;44(2):193-6. doi: 10.4103/0253-7613.93847. PMID 22529474
- [Background] Zollei E, Bertalan V, Nemeth A, Csabi P, Laszlo I, Kaszaki J, Rudas L. Non-invasive detection of hypovolemia or fluid responsiveness in spontaneously breathing subjects. BMC Anesthesiol. 2013 Nov 5;13(1):40. doi: 10.1186/1471-2253-13-40. PMID 24188480
- [Background] Tulli G. Pulse pressure variation and stroke volume variation for prediction of fluid responsiveness in critically ill patients. Crit Care Med. 2013 Jan;41(1):e11. doi: 10.1097/CCM.0b013e318270e5a1. No abstract available. PMID 23269163
- [Background] Monge Garcia MI, Gil Cano A, Gracia Romero M, Monterroso Pintado R, Perez Madueno V, Diaz Monrove JC. Non-invasive assessment of fluid responsiveness by changes in partial end-tidal CO2 pressure during a passive leg-raising maneuver. Ann Intensive Care. 2012 Mar 26;2:9. doi: 10.1186/2110-5820-2-9. PMID 22449292
- [Background] Cherpanath TG, Geerts BF, Lagrand WK, Schultz MJ, Groeneveld AB. Basic concepts of fluid responsiveness. Neth Heart J. 2013 Dec;21(12):530-6. doi: 10.1007/s12471-013-0487-7. PMID 24170232
- [Background] Vieillard-Baron A, Chergui K, Rabiller A, Peyrouset O, Page B, Beauchet A, Jardin F. Superior vena caval collapsibility as a gauge of volume status in ventilated septic patients. Intensive Care Med. 2004 Sep;30(9):1734-9. doi: 10.1007/s00134-004-2361-y. Epub 2004 Jun 26. PMID 15375649
- [Background] Pinsky MR, Payen D. Functional hemodynamic monitoring. Crit Care. 2005;9(6):566-72. doi: 10.1186/cc3927. Epub 2005 Nov 22. PMID 16356240
- [Background] Lamia B, Ochagavia A, Monnet X, Chemla D, Richard C, Teboul JL. Echocardiographic prediction of volume responsiveness in critically ill patients with spontaneously breathing activity. Intensive Care Med. 2007 Jul;33(7):1125-1132. doi: 10.1007/s00134-007-0646-7. Epub 2007 May 17. PMID 17508199
- [Background] Muller L, Bobbia X, Toumi M, Louart G, Molinari N, Ragonnet B, Quintard H, Leone M, Zoric L, Lefrant JY; AzuRea group. Respiratory variations of inferior vena cava diameter to predict fluid responsiveness in spontaneously breathing patients with acute circulatory failure: need for a cautious use. Crit Care. 2012 Oct 8;16(5):R188. doi: 10.1186/cc11672. PMID 23043910
- [Background] Jabalameli M, Soltani HA, Hashemi J, Behdad S, Soleimani B. Prevention of post-spinal hypotension using crystalloid, colloid and ephedrine with three different combinations: A double blind randomized study. Adv Biomed Res. 2012;1:36. doi: 10.4103/2277-9175.100129. Epub 2012 Aug 28. PMID 23326767
- [Background] Buggy DJ, Power CK, Meeke R, O'Callaghan S, Moran C, O'Brien GT. Prevention of spinal anaesthesia-induced hypotension in the elderly: i.m. methoxamine or combined hetastarch and crystalloid. Br J Anaesth. 1998 Feb;80(2):199-203. doi: 10.1093/bja/80.2.199. PMID 9602585
- [Background] Zhang Z, Xu X, Ye S, Xu L. Ultrasonographic measurement of the respiratory variation in the inferior vena cava diameter is predictive of fluid responsiveness in critically ill patients: systematic review and meta-analysis. Ultrasound Med Biol. 2014 May;40(5):845-53. doi: 10.1016/j.ultrasmedbio.2013.12.010. Epub 2014 Feb 2. PMID 24495437
- [Background] Bodson L, Vieillard-Baron A. Respiratory variation in inferior vena cava diameter: surrogate of central venous pressure or parameter of fluid responsiveness? Let the physiology reply. Crit Care. 2012 Nov 28;16(6):181. doi: 10.1186/cc11824. PMID 23185986
- [Background] Schmidt GA, Kory P. Ultrasound-guided central venous catheter insertion: teaching and learning. Intensive Care Med. 2014 Jan;40(1):111-3. doi: 10.1007/s00134-013-3093-7. Epub 2013 Sep 7. No abstract available. PMID 24013437
- [Background] Carpenter RL, Caplan RA, Brown DL, Stephenson C, Wu R. Incidence and risk factors for side effects of spinal anesthesia. Anesthesiology. 1992 Jun;76(6):906-16. doi: 10.1097/00000542-199206000-00006. PMID 1599111
- [Background] Marik PE. Techniques for assessment of intravascular volume in critically ill patients. J Intensive Care Med. 2009 Sep-Oct;24(5):329-37. doi: 10.1177/0885066609340640. PMID 19648183
- [Background] Funk DJ, Moretti EW, Gan TJ. Minimally invasive cardiac output monitoring in the perioperative setting. Anesth Analg. 2009 Mar;108(3):887-97. doi: 10.1213/ane.0b013e31818ffd99. PMID 19224798
- [Background] Barbier C, Loubieres Y, Schmit C, Hayon J, Ricome JL, Jardin F, Vieillard-Baron A. Respiratory changes in inferior vena cava diameter are helpful in predicting fluid responsiveness in ventilated septic patients. Intensive Care Med. 2004 Sep;30(9):1740-6. doi: 10.1007/s00134-004-2259-8. Epub 2004 Mar 18. PMID 15034650
- [Derived] Ceruti S, Minotti B, De Vivo S, De Christophoris P, Anselmi L, Saporito A. PROtocolized care to reduce HYpotension after spinal anaesthesia (ProCRHYSA randomized trial): Study protocol for a randomized controlled trial. Contemp Clin Trials Commun. 2016 Jun 29;4:39-45. doi: 10.1016/j.conctc.2016.06.012. eCollection 2016 Dec 15. PMID 29736468
- See also: Swiss Ethic — https://www.swissethics.ch/it/
- See also: Cantonal Ethic Committee — https://www4.ti.ch/dss/dsp/us/ce/comitato/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All consecutive patient undergone spinal anesthesia
Pre-assignment Details: Study began at the arrival in the operating block and ended 30 minutes after completion of spinal anaesthesia. The pre-anaesthetic phase running from time 0 to the beginning of spinal anaesthesia, the anaesthetic phase which corresponds to spinal anaesthesia gesture, followed by the post-anaesthetic phase ending 30 minutes spinal anaesthesia
Groups:
- Trans-Thoracic Echocardiography: In addition to the current clinical standard (arm A of the study) a trans-thoracic echocardiography is performed with the aim of assessing patient's volume status, identifying if he is responsive to fluid and could benefit from their administration. The echocardiography is performed with the subcostal projection to assess the size of the abdominal inferior vena cava and its collapsing during breathing.
  According to different pre-established parameters, the patient is defined as unresponsive to fluids or responsive. If it's not responsive, he proceed to spinal anesthesia. Otherwise investigators proceed to the administration of crystalloid (NaCl 0.9% or Hartmann's solution second clinical evaluation) and at the end he's rerun an echocardiographic assessment.
  Trans-thoracic echocardiography: Subcostal evaluation of inferior vena cava dimensions and colorability with cyclic spontaneous breathing in order to determine if the patients will be fluid responsive or not.
- Passive Leg Raising Test: In addition to the arm A of the study, is performed a measurement of systemic pressure with a patient positioned in semi-recumbent position. After, investigators run the Passive Leg Raising Test (PLRT): the position of the bed is changed in such manner to bring the trunk from 45° to 0° and accordingly the legs from 0° to 45°. Measurements are performed before and during the maneuver (at one minute): an increase of 5% of the systolic blood pressure is interpreted as a responsiveness to liquids.
  If the patient is not responsive to fluids, the patient is moving to the spinal anesthesia. If the patient is responsive investigators proceed to bolus administration, the patient returns to the initial PLRT position and is run again the PLRT until the patient is no longer responsive to fluids.
  Passive Leg Raising Test: Application of this test in a standard manner in order to determine if our spontaneous breathing patients are fluid responsive before spinal anesthesia.
Period: Overall Study
Arm/Group | Standard Clinical Practice | Trans-Thoracic Echocardiography | Passive Leg Raising Test
Started | 149 | 132 | 148
Completed | 149 | 132 | 148
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Clinical Practice | Trans-Thoracic Echocardiography | Passive Leg Raising Test | Total
Number analyzed (Participants) | 149 | 132 | 148 | 429
Age, Categorical [Count of Participants; unit: Participants] — Population: This analysis was intended as per-protocol analysis
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 87 | 80 | 88 | 255
    >=65 years | 62 | 52 | 60 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: This analysis was intended as per-protocol analysis
  years | 58.7 (18.0) | 55.9 (18.3) | 57.2 (18.8) | 57.2 (18.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This analysis was intended as per-protocol analysis
  Participants
    Female | 59 | 50 | 57 | 166
    Male | 90 | 82 | 91 | 263
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: This analysis was intended as per-protocol analysis
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 149 | 132 | 148 | 429
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland | 149 | 132 | 148 | 429

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Systemic Hypotensions
Description: Primary objective is to quantify significant hypotension rate after spinal anesthesia in patients brought to euvolemia according to the Trans-Thoracic Echocardiography and PLRT (Passive Leg Raising Test), compared to patients treated with the current standard. For arterial hypotension, in accordance with the international standard definitions, now define a drop in systolic blood pressure over 50 mmHg from baseline, an absolute value of systolic blood pressure less than 80 mm Hg, a mean arterial pressure below 60 mmHg or hypotension clinically symptomatic (dizziness, pallor, sweating, nausea).
Time Frame: 30 minutes
Population: Participants with Systemic Hypotensions
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: This arm is considered the current clinical standard for spinal anesthesia; its used as a control sample and statistical reference. During the induction phase the patient is fitted with a non-invasive blood pressure monitoring, three-lead ECG, pulse oximetry and peripheral intravenous device. The pressure control is set as the standard every 5 minutes until the procedure under spinal anesthesia, the cuff pressure is placed on the arm that is going to be on top during spinal anesthesia.
  Data is recorded and vital signs of the patient and is put an infusion of crystalloid (0.9% NaCl or Ringer's acetate) with administration of 500 ml during the entire procedure until the beginning of the operation.
- Arm B: In addition to the current clinical standard (arm A of the study) a trans-thoracic echocardiography is performed with the aim of assessing patient's volume status, identifying if he is responsive to fluid and could benefit from their administration. The echocardiography is performed with the subcostal projection to assess the size of the abdominal inferior vena cava and its collapsing during breathing.
  According to different pre-established parameters, the patient is defined as unresponsive to fluids or responsive. If it's not responsive, he proceed to spinal anesthesia. Otherwise investigators proceed to the administration of crystalloid (NaCl 0.9% or Hartmann's solution second clinical evaluation) and at the end he's rerun an echocardiographic assessment.
  Trans-thoracic echocardiography: Subcostal evaluation of inferior vena cava dimensions and colorability with cyclic spontaneous breathing in order to determine if the patients will be fluid responsive or not.
- Arm C: In addition to the arm A of the study, is performed a measurement of systemic pressure with a patient positioned in semi-recumbent position. After, investigators run the Passive Leg Raising Test (PLRT): the position of the bed is changed in such manner to bring the trunk from 45° to 0° and accordingly the legs from 0° to 45°. Measurements are performed before and during the maneuver (at one minute): an increase of 5% of the systolic blood pressure is interpreted as a responsiveness to liquids.
  If the patient is not responsive to fluids, the patient is moving to the spinal anesthesia. If the patient is responsive investigators proceed to bolus administration, the patient returns to the initial PLRT position and is run again the PLRT until the patient is no longer responsive to fluids.
  Passive Leg Raising Test: Application of this test in a standard manner in order to determine if our spontaneous breathing patients are fluid responsive before spinal anesthesia.
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 149 | 132 | 148
Participants | 68 | 46 | 65

2. Secondary Outcome: Pre-anesthesia Fluid Amount
Description: A secondary objective is to quantify the water administration among the three comparison groups before spinal anesthesia, using the patients in the control group as a reference, in order to assess whether these techniques are associated with more fluid administration.
Time Frame: Time between operating room entry and spinal anesthesia, up to 30 min.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 149 | 132 | 148
ml | 141 (135) | 336 (314) | 168 (237)

3. Secondary Outcome: Post-anesthesia Fluid Amount
Description: Another secondary objective is to quantify the water administration among the three comparison groups after spinal anesthesia, using the patients in the control group as a reference, in order to assess whether the techniques of filling, titrate echocardiographic evaluations and/or response to the mobilization of internal liquids are associated with lower dose, does not require more liquid.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 149 | 132 | 148
ml | 312 (424) | 257 (266) | 342 (321)

ADVERSE EVENTS:
Time Frame: Severe adverse events were measured during all surgical procedure just after the anesthesia (30 minutes).
Arm/Group | Standard Clinical Practice | Trans-Thoracic Echocardiography | Passive Leg Raising Test
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/132 | 0/148
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/132 | 0/148
Other Adverse Events (participants affected / at risk) | 1/149 | 0/132 | 0/148
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Clinical Practice (N=149) | Trans-Thoracic Echocardiography (N=132) | Passive Leg Raising Test (N=148)
Vancomycine allergy (Immune system disorders) | 1 | 0 | 0 — Cutaneous rash during Vancomycine administration

LIMITATIONS AND CAVEATS:
* single-centre study
* impossible to blind patients about their group allocation
* ultrasounds could be not feasible in a certain amount of patients due to poor ultrasound windows
* we included only American Society Anesthesiology I-III patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT02070276/Prot_SAP_000.pdf